CLINICAL TRIAL: NCT04308109
Title: Simulation Training in the Pediatric Tracheostomy and Home Ventilator Population
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Children's Wisconsin (Unknown)
Responsible Party: Principal Investigator, Jennifer Henningfeld, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 979984
Record Dates: First submitted 2019-12-16; First posted 2020-03-13 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Tracheostomy Complication; Simulation of Physical Illness; Teach-Back Communication
Keywords: Simulation; Teach-back; Caregiver
MeSH Terms: conditions — Teach-Back Communication

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): No intervention, the same as the current state of education. Caregivers will still complete the teaching and post-discharge surveys (QDTS and PDCDS) and be followed for a year after discharge.
- Active study (Experimental): In addition to the current state of education, the active study group will undergo highly realistic simulation. This involves the use of a highly realistic tracheostomy mannequin and audiovisual devices which will be used to replicate emergent clinical situations. If home invasive ventilation is anticipated, a home ventilator will be used. Caregivers will complete the teaching and post-discharge surveys (QDTS and PDCDS) and be followed for a year after discharge.
  Interventions: Behavioral: Simulation
- Active control (Active Comparator): In addition to the current state of education, the active control will undergo low-fidelity simulation that approximates the highly realistic clinical scenarios except with the use of a low-fidelity doll equipped with a tracheostomy and without the audiovisual inputs. If home invasive ventilation is anticipated, a home ventilator will be used. Caregivers still complete the teaching and post-discharge surveys (QDTS and PDCDS) and be followed for a year after discharge.
  Interventions: Behavioral: Simulation

INTERVENTIONS:
Behavioral: Simulation — Simulation involves the use of a highly realistic tracheostomy mannequin and audiovisual devices which will be used to replicate emergent clinical situations. If home invasive ventilation is anticipated, a home ventilator will be used. The simulation will last approximately 2 hours and will end with reviewing the taped session as part of debriefing. Both active arms will occur in the simulation center or sleep lab and replicate the same clinical situations by the same simulation instructor.
  Arms: Active control; Active study

SUMMARY:
The investigators will develop, refine and pilot a highly-realistic simulation program that will allow caregivers opportunities to manage critical situations as it pertains to a medically complex child dependent on tracheostomy with or without home ventilation. The investigators hope to demonstrate that the use of highly realistic simulation training will improve hospital utilization as caregivers will have a more realistic understanding of clinical and equipment-related emergencies that may occur outpatient.

DETAILED DESCRIPTION:
The investigators propose a prospective randomized control trial evaluating the use of simulation to prepare caregivers for the discharge of children dependent on respiratory technology. All caregivers of children who are (1) inpatient with a newly placed tracheostomy tube and (2) anticipated to start discharge teaching after the first date of Institutional Review Board (IRB) approval will be enrolled, regardless of home ventilator need. Caregivers with prior experience caring for tracheostomies within the last 10 years will be excluded. Estimated sample size is 60 caregivers (trainees) (2 trained caregivers anticipated per child). Trainees must be able to speak and read English.

All trainees will be randomized by child (up to 4 per child) into one of three arms (Figure 1), stratified by the need for invasive home ventilation and randomized in blocks of four. All trainees will complete our current state of education including bedside education provided by Pediatric Intensive Care Unit (PICU) or Neonatal Intensive Care Unit (NICU) nursing staff and a formal classroom-based skills class (either a 'tracheostomy-only' or a 'tracheostomy/home ventilator' class) taught by a Children's Hospital of Wisconsin (CHW) Tracheostomy and Home Ventilator respiratory therapist or durable medical equipment company (DME) respiratory therapist, and an individual scenario-based review of equipment and skills workshop with a CHW Tracheostomy and Home Ventilator Respiratory Therapist.

In addition to the current state of education, the active study group will also undergo highly realistic simulation. This involves the use of a highly realistic tracheostomy mannequin and audiovisual devices which will be used to replicate emergent clinical situations. If home invasive ventilation is anticipated, a home ventilator will be used. The active control will undergo low-fidelity simulation that approximates the highly realistic clinical scenarios except with the use of a low-fidelity doll equipped with a tracheostomy and without the audiovisual inputs. Both active arms will occur in the simulation center or sleep lab and replicate the same clinical situations by the simulation instructor. After the simulation, participants will be debriefed by the instructor, who will use a tape of their session as a teaching tool.

Commonly encountered emergent outpatient problems to be simulated include 1) obstructed tracheostomy tube leading to the need for cardiopulmonary resuscitation; 2) bleeding from the tracheostomy tube; 3) acute desaturation and/or bradycardia; and 4) accidental decannulation. If invasive home ventilation is anticipated, ventilator alarm troubleshooting for high pressure alarms, low minute ventilation alarms, auto-cycling of the ventilator and water in the tubing will be included in the simulation.

All trainees will undergo a teach-back session with a CHW Tracheostomy and Home Ventilator Program respiratory therapist during which essential skills and responses to clinical situations are assessed. If a trainee passes this session, the respiratory therapist has determined that they have met criteria to move onto independent care sessions and the trainees have acquired the trach and home ventilator knowledge to provide care in the home. If a trainee fails this teach-back session, the information failed will be reviewed and the family will repeat the teach-back session until they pass and then move into independent care sessions. Independent care sessions are practical demonstrations of all skills needed to take care of the child at home. Independent care sessions are repeated until all skills have been passed. Teach-back and independent care sessions are part of the current state of education.

ELIGIBILITY:
Anticipated count of 90 participants includes 30 patients and 60 caregivers (2 per patient). Caregivers are the primary subjects, and patients are enrolled so the investigators can use their medical records.

Caregivers:

Inclusion Criteria

* Must be able to read and speak English
* Caring for a patient with a tracheostomy being discharged from the NICU/PICU for the first time

Exclusion Criteria

- Can not have cared for a child with a tracheostomy in the last 10 years

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2026-08-25 (Estimated); Study Completion 2026-08-25 (Estimated)

PRIMARY OUTCOMES:
Teach-back session performance | Within 4 weeks of hospital discharge
  Difference in Teach-back performance between active study and control groups. Measured from 0-24, with higher scores being better.
Independent Care session performance | Within 4 weeks of hospital discharge
  Independent Care performance between active study and control groups.
Hospital length of stay | First teaching session to discharge, an average of 4 weeks
  Difference in hospital length of stay between active study and active control groups. Measured from 0-7, with higher scores being better.
Phone Calls | 1 year after initial discharge
  Difference in number of Phone Calls (from participants to medical providers/home care company) between active and control groups.
Number of Hospital Re-admissions/Emergency Room (ER) visits | 1 year after initial discharge
  Difference in the number of Hospital Re-admissions/ER visit counts between active and control groups.

SECONDARY OUTCOMES:
Quality of discharge teaching scores | Within 48 hours of initial hospital discharge
  Quality of Discharge Teaching Scale measured on day of discharge; scale of 0 to 10; very high/very low scores indicate stronger opinions
Caregiver post-discharge coping scores | Scale administered 24 hours after discharge and about 1 month after discharge
  Post Discharge Coping Difficulty Scale administered 24 hours after discharge and at first Tracheostomy/Home Ventilator clinic visit; scale of 0 to 10; very high/very low scores indicate stronger opinions

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Henningfeld, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Wauwatosa, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No